CLINICAL TRIAL: NCT05409573
Title: Feasibility of End-tidal Oxygen Concentration Monitoring During Preoxygenation for Intubation in the Intensive Care Unit. First Part, Preliminary Study of the IMPROVE Global Project
Brief Title: Feasibility of End-tidal Oxygen Concentration Monitoring During Preoxygenation for Intubation in the Intensive Care Unit.
Acronym: IMPROVE-Pre
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHRO-2021-08
Record Dates: First submitted 2022-05-12; First posted 2022-06-08 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Critically Ill
Keywords: Preoxygenation; intubation; end-tidal of oxygen; intensive care unit; critically ill patients
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Non-comparative prospective interventional study
Masking Description: The clinician and caregivers in charge of the patient during the intubation procedure will be blinded: the facemask EtO2 and pharyngeal EtO2 will not be visible on the monitor for them
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- monitoring of the expired oxygen fraction (Experimental): A double monitoring of EtO2 will be performed during the procedure of intubation (from the beginning of the preoxygenation to the success of intubation):
  * In the pharynx (via a nasopharyngeal catheter) for the needs of the study
  * On the facemask (as the practice in the OR)
  Interventions: Other: double monitoring of EtO2

INTERVENTIONS:
Other: double monitoring of EtO2 — A double monitoring of EtO2 will be performed during the procedure of intubation (from the beginning of the preoxygenation to the success of intubation):
  * In the pharynx (via a nasopharyngeal catheter) for the needs of the study
  * On the facemask (as the practice in the OR)

SUMMARY:
Intubation is a common procedure in the intensive care unit. Hypoxemia is the most frequent complication of this procedure.

Monitoring the end-tidal of oxygen is recommended in operating room (OR). End-tidal of oxygen (EtO2) >90% is an indication of a correct preoxygenation.

This monitoring is not used in routine in intensive care unit (ICU). There is no recommendation on the monitoring of end-tidal of oxygen in intensive care unit. In practice, clinicians use pulsed oxygen saturation (SpO2) to determine whether the patient is sufficiently preoxygenated. However, this parameter is not a good indicator of a correct preoxygenation.

In the OR, patients are compliant during the preoxygenation period and the measure of EtO2 with the face mask monitor is considered reliable because i) mask leakage is minimal and ii) the patient can breathe slowly and regularly.

Theses conditions are not available in critical ill patients requiring emergency intubation. EtO2 measured on the facemask may not reflect true EtO2.

This concern about the reliability of EtO2 measurement via the facemask justifies that we conduct a study to compare EtO2 measured on a facemask (facemask EtO2) to EtO2 measured in pharynx (via e nasopharyngeal catheter).

The aim of this study is to determine whether the measurement of EtO2 on facemask is reliable in patients in ICU.

DETAILED DESCRIPTION:
This is a prospective non-comparative interventional study.

A double monitoring of EtO2 will be performed during the procedure of intubation (from the beginning of the preoxygenation to the success of intubation):

* In the pharynx (via a nasopharyngeal catheter) for the needs of the study
* On the facemask (as the practice in the OR) The duration of the study will not exceed one hour, including the installation of the devices.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Requiring an intubation in ICU for acute respiratory failure defined as a respiratory rate ≥ 25/min or clinical signs of respiratory distress or hypoxemia defined as oxygen requirement ≥ 15L/min or FiO2 ≥80% to maintain SpO2 ≥92% or a PaO2/FiO2 ratio <100 mmHg
* With preoxygenation by noninvasive ventilation

Exclusion Criteria:

* Intubation for cardiac arrest
* EtO2 monitoring not available
* Pulsed oxygen saturation monitoring specific for the study not available
* Preoxygenation by high-flow nasal oxygen therapy or bag-mask ventilation
* Allergy to lidocaine (for local nasal anesthesia)
* Previously
* Patient not affiliated or excluded from social protection, or under law protection (namely minors, pregnant or breastfeeding women, persons deprived of their liberty by court or administrative decision)
* Previously included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-23 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of expired O2 at facemask during preoxygenation | Hour 1
  compare facemask EtO2 to pharyngeal EtO2 during preoxygenation in order to know if facemask monitoring is sufficient or if a nasopharyngeal catheter is absolutely necessary to monitor alveolar oxygenation.
Percentage of expired pharyngeal O2 during preoxygenation | Hour 1
  compare facemask EtO2 to pharyngeal EtO2 during preoxygenation in order to know if facemask monitoring is sufficient or if a nasopharyngeal catheter is absolutely necessary to monitor alveolar oxygenation.

SECONDARY OUTCOMES:
Number of patient who had a pulsed oxygen saturation under 90% | Hour 1
  Hypoxemia is defined as the occurrence of a pulsed oxygen saturation (SpO2) ≤ 90%. The end of preoxygenation is defined by the induction of anesthetics drugs. Successful intubation is defined by the presence of 3 identical waveforms on the capnograph.

CONTACTS AND LOCATIONS:
Overall Officials: Mai-Anh NAY, PH, Principal Investigator — CHR d'Orléans
Locations (1):
- CHR d'ORLEANS, Orléans, France

REFERENCES:
- [Background] Carrillo A, Gonzalez-Diaz G, Ferrer M, Martinez-Quintana ME, Lopez-Martinez A, Llamas N, Alcazar M, Torres A. Non-invasive ventilation in community-acquired pneumonia and severe acute respiratory failure. Intensive Care Med. 2012 Mar;38(3):458-66. doi: 10.1007/s00134-012-2475-6. Epub 2012 Feb 9. PMID 22318634
- [Background] Thille AW, Frat JP, Brun-Buisson C. Trends in use and benefits of non-invasive ventilation as first-line therapy in acute respiratory failure. Intensive Care Med. 2014 Aug;40(8):1179-80. doi: 10.1007/s00134-014-3370-0. Epub 2014 Jun 25. No abstract available. PMID 24962719
- [Background] Ozsancak Ugurlu A, Sidhom SS, Khodabandeh A, Ieong M, Mohr C, Lin DY, Buchwald I, Bahhady I, Wengryn J, Maheshwari V, Hill NS. Use and outcomes of noninvasive positive pressure ventilation in acute care hospitals in Massachusetts. Chest. 2014 May;145(5):964-971. doi: 10.1378/chest.13-1707. PMID 24480997
- [Background] Frat JP, Ricard JD, Quenot JP, Pichon N, Demoule A, Forel JM, Mira JP, Coudroy R, Berquier G, Voisin B, Colin G, Pons B, Danin PE, Devaquet J, Prat G, Clere-Jehl R, Petitpas F, Vivier E, Razazi K, Nay MA, Souday V, Dellamonica J, Argaud L, Ehrmann S, Gibelin A, Girault C, Andreu P, Vignon P, Dangers L, Ragot S, Thille AW; FLORALI-2 study group; REVA network. Non-invasive ventilation versus high-flow nasal cannula oxygen therapy with apnoeic oxygenation for preoxygenation before intubation of patients with acute hypoxaemic respiratory failure: a randomised, multicentre, open-label trial. Lancet Respir Med. 2019 Apr;7(4):303-312. doi: 10.1016/S2213-2600(19)30048-7. Epub 2019 Mar 18. PMID 30898520
- [Background] Jaber S, Amraoui J, Lefrant JY, Arich C, Cohendy R, Landreau L, Calvet Y, Capdevila X, Mahamat A, Eledjam JJ. Clinical practice and risk factors for immediate complications of endotracheal intubation in the intensive care unit: a prospective, multiple-center study. Crit Care Med. 2006 Sep;34(9):2355-61. doi: 10.1097/01.CCM.0000233879.58720.87. PMID 16850003